CLINICAL TRIAL: NCT05872516
Title: A Study to Evaluate Accuracy and Validity of the Chang Gung Atrial Fibrillation Detecting Software
Brief Title: Atrial Fibrillation Detecting Software Gung Atrial Fibrillation Detecting Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202200717A3
Record Dates: First submitted 2023-05-04; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Atrial Fibrillation
Keywords: artificial intelligence
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Software diagnosis (Experimental): Software diagnosis with gold standard of 3 doctors' consensus.
  Interventions: Device: Chang Gung Atrial Fibrillation Detecting Software

INTERVENTIONS:
Device: Chang Gung Atrial Fibrillation Detecting Software — This software is expected to be used in clinical testing to interpret the static 12-lead ECG of adults who are over 20 years old and suspected of having atrial fibrillation, detect whether there is a signal of atrial fibrillation, and output the results for clinicians Near-instant auxiliary diagnostic use.

SUMMARY:
Chang Gung Atrial Fibrillation Detection Software is an artificial intelligence electrocardiogram signal analysis software that detects whether a patient has atrial fibrillation by static 12-lead ECG signals. This study is a non-inferiority test based on the control group. The main purpose is to verify whether Chang Gung atrial fibrillation detection software can correctly identify atrial fibrillation in patients with atrial fibrillation, and can be used to provide a reference for doctors to detect atrial fibrillation.

DETAILED DESCRIPTION:
This study is a retrospective study, and the data is from the six hospitals of Chang Gung Medical Research Database (CGRD). We collected de-identified static 12-lead electrocardiogram (ECG) data from the database during the period of January 1, 2006, to December 31, 2019.

We created a training set and a testing set of ECG data from the CGRD. Then, we stratified and sampled ECG signals from the testing set according to the actual proportion to obtain the experimental sample.

The computer first preliminarily screened and selected ECG data that met the inclusion and exclusion criteria, and then numbered them sequentially. A cardiologist confirmed that the sampled ECG data did not include exclusion criteria.

The ECG data were converted into images and interpreted for the presence or absence of atrial fibrillation by three cardiologists. Their results were used as the gold standard (reference) for this study.

After determining the experimental standards, the ECG signals were inputted into the Chang Gung Atrial Fibrillation Detection software for analysis and interpretation of each ECG data.

After the software interpretation was completed, the results were compared with the interpretations of the physicians, and the primary and secondary evaluation indicators were analyzed accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Equal or greater than twenty years old
* Static 12-lead electrocardiogram of General Electric MUSE XML format file.
* The data comes from the static 12-lead electrocardiogram device of General Electric (model MAC5500).
* The electrocardiogram signal is 500 Hz.
* The Alternating current (AC) filter of the electrocardiogram signal is 60 Hz.

Exclusion Criteria:

* Cases used in the model development process.
* Lacks any electrode.
* Contain any electrode lacks a segment.
* Misplaced leads

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 788 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity | baseline
  The rate of test results that correctly indicate the presence.

SECONDARY OUTCOMES:
Specificity | baseline
  The rate of test results that correctly indicate the absence.
Accuracy | baseline
  The rate of all test results that correctly indicate.
Area Under the receiver operating characteristic Curve | baseline
  A graphical plot that illustrates the diagnostic ability of a binary classifier system as its discrimination threshold is varied.
Positive predictive value | baseline
  The proportions of positive results in statistics and diagnostic tests that are true positive results
Negative predictive value | baseline
  The proportions of negative results in statistics and diagnostic tests that are true negative results
False positive rate | baseline
  The rate of test result which wrongly indicates that a particular condition or attribute is present
False negative rate | baseline
  The rate of test result which wrongly indicates that a particular condition or attribute is absent

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Fu Kuo, MD/Ph.D, Study Chair — Associate Professor and Director Division of Rheumatology
Locations (1):
- Chang Gung memorial hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mant J, Fitzmaurice DA, Hobbs FD, Jowett S, Murray ET, Holder R, Davies M, Lip GY. Accuracy of diagnosing atrial fibrillation on electrocardiogram by primary care practitioners and interpretative diagnostic software: analysis of data from screening for atrial fibrillation in the elderly (SAFE) trial. BMJ. 2007 Aug 25;335(7616):380. doi: 10.1136/bmj.39227.551713.AE. Epub 2007 Jun 29. PMID 17604299
- [Background] US Preventive Services Task Force; Curry SJ, Krist AH, Owens DK, Barry MJ, Caughey AB, Davidson KW, Doubeni CA, Epling JW Jr, Kemper AR, Kubik M, Landefeld CS, Mangione CM, Silverstein M, Simon MA, Tseng CW, Wong JB. Screening for Atrial Fibrillation With Electrocardiography: US Preventive Services Task Force Recommendation Statement. JAMA. 2018 Aug 7;320(5):478-484. doi: 10.1001/jama.2018.10321. PMID 30088016
- [Background] Wong KC, Klimis H, Lowres N, von Huben A, Marschner S, Chow CK. Diagnostic accuracy of handheld electrocardiogram devices in detecting atrial fibrillation in adults in community versus hospital settings: a systematic review and meta-analysis. Heart. 2020 Aug;106(16):1211-1217. doi: 10.1136/heartjnl-2020-316611. Epub 2020 May 11. PMID 32393588
- [Background] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomstrom-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. No abstract available. PMID 32860505